CLINICAL TRIAL: NCT03391115
Title: Personalized Experiences to Inform Improved Communication for Minorities With Life Limiting Illness
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-1885.cc; 1K99NR016686-01A1 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2018-01-05 (Actual); Results first posted 2019-12-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: COPD; Heart Failure; Cancer
Keywords: Psychosocial; Underserved; Palliative; Electronic Health Record; Narrative
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Neoplasms; Narration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatient Participants: Patients admitted to University of Colorado Hospital with at least one of the following diagnoses:
  * Heart Failure
  * COPD
  * Cancer
  Interventions: Behavioral: Storytelling Intervention for Patient Participants
- Nurse Participants: Bedside nurses who provide care at the inpatient level for the following diseases:
  * Heart Failure
  * COPD
  * Cancer
  Interventions: Behavioral: Storytelling Intervention for Nurse Participants

INTERVENTIONS:
Behavioral: Storytelling Intervention for Patient Participants — The storytelling intervention consists of an audio-recorded interview with each patient participant prompted the participant to share their story with questions such as: tell me about your illness, tell me how your illness has affected your emotions, relationships, and spirituality. The interview transcripts will be used to co-create a 1 page patient story using these criteria:1) written in the first person; 2) nonjudgmental; 3) captures the participant's voice; 4) accurately reflects content of the interview; and 5) non-labeling. Once the story has been approved by the participant, I will upload it to the EHR.
  Groups: Inpatient Participants
Behavioral: Storytelling Intervention for Nurse Participants — Once the patient's story is uploaded to the EHR, automatic alerts will be sent to the participant's EHR-assigned nurses. For usability testing, nurse participants will 1) provide content expertise of the workflow processes, and 2) put the storytelling intervention through in-house usability testing to check the "strength" of EHR features and user-friendliness. Data will be collected with exit interviews and completion of a questionnaire: the System Usability Scale which asks them to rank their satisfaction with specific elements such as: how the story is labeled and presented in the EHR, any technical navigation EHR difficulties, and use of the material.
  Groups: Nurse Participants

SUMMARY:
The purpose of this research is to develop patient-centered palliative care interventions to improve patient-provider communication and Quality of Life (QoL) of ethnic and racial minority patients living with life-limiting illnesses. Eliciting personal experiences is an effective way for patients to communicate their cultural values and beliefs. This study will assess how to integrate the patients' personal experience narratives into the electronic health record (EHR). The primary hypothesis is that the implementation of a patient-centered intervention to elicit personal experiences that are included in the EHR will improve patient-provider communication and patients' QoL.

DETAILED DESCRIPTION:
Racial and ethnic minority patients with a Life Limiting Illnes (LLI) in the United States are underserved in many ways, including quality of palliative care. Specific disparities have been reported in palliative care for minority patients, including sub-optimal patient-provider communication and resulting lower QoL. A potential approach to improve communication is to elicit patients' personal narratives that address their cultural or spiritual values and beliefs, and include them in the EHR. The objective of this observational study is to assess the feasibility and efficacy of a palliative care nursing intervention designed to 1) identify barriers and facilitators for eliciting and recording relevant narratives from the perspectives of the key stakeholders: minority patients with LLI; 2) to conduct usability testing, applying a user-system-environment evaluation process to determine essential requirements for integration of the patient-centered narratives into the EHR; and 3) identify barriers and facilitators of integration of the patient's narrative into daily workflow from the perspectives of key stakeholders: acute care bedside nurse.

ELIGIBILITY:
Inclusion Criteria: Patients

* 18 years of age or older
* able to read English
* capable of giving informed consent
* self-identifying as part of a racial or ethnic minority
* diagnosed with at least one LLI. The operational definition of LLI eligible for this study includes the following diagnoses:

  1. metastatic solid cancer or inoperable lung cancer;
  2. COPD with FEV1 values < 35% predicted or oxygen dependence;
  3. New York Heart Association Class III or IV heart failure (CHF).

Inclusion criteria: Nurse

* 18 years of age or older
* Confirm verbally that they were involved in the care of a patient who is participating in the storytelling intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatient population description:
  Patient's on inpatient with the following diagnoses:
  * COPD
  * Heart Failure
  * Cancer
  Nurse patient population:
  Bedside nurses who are involved in the care of a patient who is participating in the storytelling intervention with the diagnoses listed above.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coats H, Meek PM, Schilling LM, Akard TF, Doorenbos AZ. "Connection": The Integration of a Person-Centered Narrative Intervention into the Electronic Health Record: An Implementation Study. J Palliat Med. 2020 Jun;23(6):785-791. doi: 10.1089/jpm.2019.0376. Epub 2020 Jan 6. PMID 31905039

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two Nurse participants in the dyadic patient-nurse enrollment were not successfully recruited.
Groups:
- Inpatient Participants: Patients admitted to University of Colorado Hospital with at least one of the following diagnoses:
  * Heart Failure
  * COPD
  * Cancer
  Storytelling Intervention for Patient Participants: The storytelling intervention consists of an audio-recorded interview with each patient participant prompted the participant to share their story with questions such as: tell me about your illness, tell me how your illness has affected your emotions, relationships, and spirituality. The interview transcripts will be used to co-create a 1 page patient story using these criteria:1) written in the first person; 2) nonjudgmental; 3) captures the participant's voice; 4) accurately reflects content of the interview; and 5) non-labeling. Once the story has been approved by the participant, I will upload it to the EHR.
- Nurse Participants: Bedside nurses who provide care at the inpatient level for the following diseases:
  * Heart Failure
  * COPD
  * Cancer
  Storytelling Intervention for Nurse Participants: Once the patient's story is uploaded to the EHR, automatic alerts will be sent to the participant's EHR-assigned nurses. For usability testing, nurse participants will 1) provide content expertise of the workflow processes, and 2) put the storytelling intervention through in-house usability testing to check the "strength" of EHR features and user-friendliness. Data will be collected with exit interviews and completion of a questionnaire: the System Usability Scale which asks them to rank their satisfaction with specific elements such as: how the story is labeled and presented in the EHR, any technical navigation EHR difficulties, and use of the material.
Period: Overall Study
Arm/Group | Inpatient Participants | Nurse Participants
Started | 20 | 18
Completed | 20 | 18 (Two Nurse participants in the dyadic patient-nurse enrollment were not successfully recruited.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inpatient Participants | Nurse Participants | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Full Range); unit: years] | 52.15 [29 to 72] | 31.39 [23 to 53] | 41.77 [23 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 12 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 0 | 9
  Not Hispanic or Latino | 11 | 18 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 0 | 11
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 0 | 17 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Completed Exit Interviews From Patients on Feasibility of Their Use of Their Narrative Integrated Into EHR
Description: Using an observational design, this measure (exit interviews) were completed with 20 inpatient participants and 18 nurse participants. The qualitative data from the interviews were used to define and refine the storytelling intervention. The data collected from the exit interview is qualitative in nature and therefore does not have a numerical value.
Time Frame: 1-2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Inpatient Participants | Nurse Participants
Number analyzed (Participants) | 20 | 18
Participants | 20 | 18

2. Other Pre Specified Outcome: Usability Assessment Via the System Usability Scale(SUS), Range of 0 to 100, With Higher Number Representing a Better Outcome SUS Scores Have a Range of 0 to 100, the Higher the Number Represents a Better Outcome.
Description: This study will utilize an observational design to define and refine the storytelling intervention, seeking input from the key stakeholders: providers (acute care bedside nurses).The SUS scale is a 10 item Likert scale which gives a global view of subjective assessment of usability with five item responses options from strongly agree to strongly disagree. SUS yields a single number representing a composite measure of the overall usability of the system being studied. Note that scores for individual items are not meaningful on their own. To calculate the SUS score, first sum the score contributions from each item. Each item's score contribution will range from 0 to 4. For items 1,3,5,7, and 9, the score contribution is the scale position minus 1. For items 2,4,6,8, and 10, the contribution is 5 minus the scale position. Multiply the sum of the scores by 2.5 to obtain the overall value of the SUS, with the higher the number, the better the outcome.
Time Frame: 1-2 weeks
Population: Patient Participants did not complete this secondary measure. This was only the nurse participants completing the NIH System Usability Scale
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Inpatient Participants | Nurse Participants
Number analyzed (Participants) | 0 | 18
score on a scale |  | 89.71 [75 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events occurred.
Arm/Group | Inpatient Participants | Nurse Participants
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT03391115/Prot_000.pdf
  • Informed Consent Form (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03391115/ICF_001.pdf